CLINICAL TRIAL: NCT03868813
Title: An Artificial Intelligence Assisted Telehealth Intervention to Promote Self-Management in Patients With Type 2 Diabetes Mellitus (Qualitative Interview)
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Mohanraj Thirumalai, Assistant Professor, University of Alabama at Birmingham
Other Study IDs: UAB-DRC-2019-1
Record Dates: First submitted 2019-03-05; First posted 2019-03-11 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Interview with People with Diabetes: One-on-One interview with people with diabetes
  Interventions: Behavioral: Semi-structured Interview
- Interview with Health Coaches: One-on-One interview with health coaches
  Interventions: Behavioral: Semi-structured Interview

INTERVENTIONS:
Behavioral: Semi-structured Interview — One-on-one semi-structured interviews

SUMMARY:
This protocol involves a qualitative study of the needs/preferences of people with diabetes and health coaches regarding a telehealth coaching platform for glycemic control in people with diabetes.

ELIGIBILITY:
Inclusion Criteria:

Health Coaches Group:

(i) age between 18 and 80 years (ii) fluent in English (iii) work in or carry expertise in physical activity, nutrition/diet or health behavior.

People with Diabetes Group (Patient/Caregiver Dyads):

(i) age between 18 and 80 years (ii) fluent in English (iii) have Type-II diabetes.

Exclusion Criteria:

None

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: There will be a total of two 2 groups - one group comprising of 10 health experts and another group 2comprising of 10 patient/caregiver dyads (20 people). There is no treatment or intervention offered, only the interview questionnaire will differ based on the group.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Users' Expectation from a Health Coaching System | 60 minutes
  This interview with participants help produce knowledge on the users' expectations from a health coaching system

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States